CLINICAL TRIAL: NCT07192627
Title: Selective Endoscopic Resection vs. Surveillance Following CRT for Rectal Cancer: 1-Year Oncologic and Functional Outcomes
Brief Title: ESD in Locally Advanced Rectal Cancer Following CRT
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Yusuf Salah-eldin Amry Ahmad, Assistent Lecturer at Tropical Medicine and Gastroenterology, Assiut University
Other Study IDs: ESD in rectal cancer
Record Dates: First submitted 2025-09-11; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Residual mucosal lesion amenable for ESD after CRT: Mucosal lesions following CRT amenable for ESD will be resected with pathological examination
  Interventions: Procedure: Endoscopic mucosal dissection
- Residual mucosal lesion not amenable for ESD after CRT: wait and watch strateagy

INTERVENTIONS:
Procedure: Endoscopic mucosal dissection — Removal of lesions extending down to submucosa
  Groups: Residual mucosal lesion amenable for ESD after CRT

SUMMARY:
residual mucosal lesions in patients with locally advanced rectal cancer after CRT are still confusing for decision to continue follow up or excise.

Investigators decided to compare two groups with cCR or nCR with MDT management decision to whether do ESD for this residual lesion or continue follow up and its effect on disease free survival.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) represents a significant health challenge in Egypt. According to GLOBOCAN 2020, rectal cancer ranks sixth in all cancers among males and females, with 5,231 new cases, accounting for 3.9% of all cancers. El-Moselhy et al., 2025 reported that the rectum was involved in up to 20% of CRC cases in Egypt .

In recent years, there was a shift in management of locally advanced rectal cancer (LARC) toward organ preserving strategies. After neoadjuvant chemoradiotherapy (CRT) or total neoadjuvant therapy (TNT), a notable proportion of patients achieve a clinical complete response (cCR) or near-complete response (nCR) making them candidates for either structured watch-and-wait (W&W) surveillance or selective local interventions designed to avoid total mesorectal excision (TME) .

In phase II OPRA trial, long-term organ preservation was achieved in approximately 50% of participants, with most tumor regrowth occurring within the first two years.

Despite that, small residual mucosal/submucosal lesions with cCR post CRT are still challenging in management with either W&W or ESD. Endoscopic submucosal dissection (ESD) offers en-bloc resection, comprehensive histopathologic evaluation (depth of invasion, lymphovascular invasion, budding, margins), and the option of salvage surgery if needed. Early evidence supports its feasibility and safety in this setting .

One meta-analysis confirms strong effectiveness and low rate of recurrence when ESD is used for residual or recurrent lesions with prior surgery or endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with rectal adenocarcinoma who underwent full course locoregional chemoradiotherapy with organ-preservation intent.

Post-CRT assessment showing either:

A. Small residual mucosal/submucosal lesion amenable to en-bloc ESD (CRT→ESD), OR B. Clinical/radiologic near-complete/complete response and decision to observe (CRT→Follow-up).

Exclusion Criteria:

* - Evidence of distant metastasis at post-CRT restaging.
* Lesions unsuitable for endoscopic resection (circumferential, deeply invasive on EUS/MRI).
* Patients who had immediate TME after CRT for other reasons.
* Unfit for endoscopy or follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who completed locoregional chemoradiotherapy with organ preservation intent will be prospectively enrolled. Post-CRT restaging at 8-12 weeks will be discussed at MDT. Patients with a small residual mucosal/submucosal lesion amenable to en-bloc endoscopic resection will be offered ESD (CRT→ESD). Patients with clinical/radiologic complete or near-complete response and no endoscopically resectable residual lesion will be managed with structured surveillance (CRT→Follow-up)
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
- Compare 1-year disease-free survival (DFS) between patients treated with ESD for small residual rectal lesions after locoregional CRT (CRT→ESD) and patients managed with close surveillance after CRT (CRT→Follow-up). | one year
  Compare 1-year disease-free survival (DFS) between patients treated with ESD for small residual rectal lesions after locoregional CRT (CRT→ESD) and patients managed with close surveillance after CRT (CRT→Follow-up)

SECONDARY OUTCOMES:
- Compare local regrowth/recurrence rates at 1 year between the two groups. - Compare organ-preservation rate at 1 year (proportion avoiding TME). | One year
  - Compare local regrowth/recurrence rates at 1 year between the two groups.
Compare organ-preservation rate at 1 year (proportion avoiding TME). | One year
  The need for surgery in either group

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

REFERENCES:
- [Background] Verheij FS, Omer DM, Williams H, Lin ST, Qin LX, Buckley JT, Thompson HM, Yuval JB, Kim JK, Dunne RF, Marcet J, Cataldo P, Polite B, Herzig DO, Liska D, Oommen S, Friel CM, Ternent C, Coveler AL, Hunt S, Gregory A, Varma MG, Bello BL, Carmichael JC, Krauss J, Gleisner A, Guillem JG, Temple L, Goodman KA, Segal NH, Cercek A, Yaeger R, Nash GM, Widmar M, Wei IH, Pappou EP, Weiser MR, Paty PB, Smith JJ, Wu AJ, Gollub MJ, Saltz LB, Garcia-Aguilar J. Long-Term Results of Organ Preservation in Patients With Rectal Adenocarcinoma Treated With Total Neoadjuvant Therapy: The Randomized Phase II OPRA Trial. J Clin Oncol. 2024 Feb 10;42(5):500-506. doi: 10.1200/JCO.23.01208. Epub 2023 Oct 26. PMID 37883738
- [Background] Leung G, Nishimura M, Hingorani N, Lin IH, Weiser MR, Garcia-Aguilar J, Pappou EP, Paty PB, Schattner MA. Technical feasibility of salvage endoscopic submucosal dissection after chemoradiation for locally advanced rectal adenocarcinoma. Gastrointest Endosc. 2022 Aug;96(2):359-367. doi: 10.1016/j.gie.2022.02.014. Epub 2022 Feb 17. PMID 35183541
- [Background] Ferlay, J., Ervik, M., Lam, F., Colombet, M., Mery, L., Piñeros, M., Znaor, A., Soerjomataram, I. & Bray, F. (2020) Global Cancer Observatory: Cancer Today. Rectum Fact Sheet. Accessed 5 September 2025 edn. Lyon, France, International Agency for Research on Cancer.
- [Background] El-Moselhy, E. A., Abdel-Halim, M. M., Eid, A. M. M. E., Ghazy, A. M., Abdelmageed, N. A., Eldamaty, A. A., Sherif, S. A., Attia, A. A., Kotb, F. M., Abdelhafez, A. A., Abdelnaser, M. M., El Sisi, M. H., Abdelnaby, A. M., Ibrahim, M. A., Khalil, O. O., Tag El-Din, M., Osman, E. M., Mohammed, A.-E. S., Abo-Rahma, A. H., Abdrabo, A. E., El Guindy, A. M. & Kholief, K. M. S. (2025) Colorectal cancer risk factors: A multi-center, case-control study in Egypt. Clinical Epidemiology and Global Health. 33. doi: 10.1016/j.cegh.2025.102017.
- [Background] Eisele M, Ceccacci A, Gupta M, Heer E, Elhanafi S, Ngamruengphong S, Thosani N, Iannuzzi J, Kumar P, Belletrutti P, Gill R, Forbes N. Effectiveness and safety of endoscopic submucosal dissection for residual or recurrent colorectal neoplasia: Meta-analysis. Endosc Int Open. 2025 Jul 1;13:a26060982. doi: 10.1055/a-2606-0982. eCollection 2025. PMID 40611847
- [Background] Dossa F, Chesney TR, Acuna SA, Baxter NN. A watch-and-wait approach for locally advanced rectal cancer after a clinical complete response following neoadjuvant chemoradiation: a systematic review and meta-analysis. Lancet Gastroenterol Hepatol. 2017 Jul;2(7):501-513. doi: 10.1016/S2468-1253(17)30074-2. Epub 2017 May 4. PMID 28479372